CLINICAL TRIAL: NCT06658964
Title: A Single-center, Non-randomized, Open-label, Self-controlled Phase 1 Clinical Study to Evaluate Drug-drug Interactions of JMKX003142 Tablets in Healthy Subjects
Brief Title: Study to Evaluate the Drug-drug Interaction of JMKX003142 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Collaborators: Zhejiang Hangyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMKX003142-102
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: ADPKD (autosomal Dominant Polycystic Kidney Disease)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1：JMKX003142 and itraconazole (Experimental): Interaction between JMKX003142 and itraconazole
  Interventions: Drug: Cohort 1: JMKX003142 and itraconazole
- Cohort 2：JMKX003142 and rifampicin (Experimental): Interaction between JMKX003142 and rifampicin
  Interventions: Drug: Cohort 2: JMKX003142 and rifampicin

INTERVENTIONS:
Drug: Cohort 1: JMKX003142 and itraconazole — JMKX003142: Dose: 3 mg, D1, once only in the morning. 3 mg JMKX003142 coadministered with 200 mg itraconazole once: Day8, once only in the morning.
  Itraconazole：Dose: 200mg once；Day5-Day7 and Day9-Day11, QD
  Arms: Cohort 1：JMKX003142 and itraconazole
Drug: Cohort 2: JMKX003142 and rifampicin — JMKX003142: Dose: 6 mg, D1, once only in the morning. 3 mg JMKX003142 coadministered with 200 mg rifampicin once: Day14, once only in the morning.
  Rifampicin：Dose: 600mg once；Day5-Day13 and Day15-Day17, QD
  Arms: Cohort 2：JMKX003142 and rifampicin

SUMMARY:
To evaluate the effects of oral administration rifampicin or itraconazole capsules on the pharmacokinetics of JMKX003142 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the research content, process, and potential risks of this trial, voluntarily participate in the clinical trial and sign the informed consent,
* Healthy male and female subjects aged ≥18 years and ≤45 years old, Male weight ≥50kg, female weight ≥45kg, body mass index ≥19 kg/m2 and ≤28 kg/m2,
* The health of the subjects was determined by the investigator based on medical history, physical examination, clinical laboratory examination, and 12-lead electrocardiogram, all of which were determined by the investigator to be normal or not clinically significant.

Exclusion Criteria:

* HBV surface antigen, HCV antibody, HIV, or syphilis are positive during screening,
* At the time of screening, the vital signs are within the following ranges: systolic blood pressure <90 mmHg or >140 mmHg, diastolic blood pressure <50 mmHg or >90 mmHg, pulse <50 bpm or >100 bpm and ear temperature 37.5℃or<35℃,
* More than 5 cigarettes per day during the 3 months prior to screening, Or were unable to quit smoking/containing tobacco products during the trial,
* Have special requirements for diet and cannot comply with the diet provided and corresponding regulations.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Cmax of JMKX003142 in plasma | approximately 5 days after JMKX003142 administered
  Cmax of JMKX003142 when JMKX003142 administered with or without itraconazole/rifampicin
AUC of JMKX003142 in plasma | approximately 5 days after JMKX003142 administered
  AUC of JMKX003142 when JMKX003142 administered with or without itraconazole/rifampicin

CONTACTS AND LOCATIONS:
Overall Officials: Leilei Zhu, Principal Investigator — Shuguang Hospital Affiliated with Shanghai University of TCM